CLINICAL TRIAL: NCT05015647
Title: Is There Any Indication for Protein Free Products in Patients With Advanced CKD at Risk of Malnutrition?A Pilot Randomized Controlled Trial
Brief Title: Low Protein Diet in CKD Patients at Risk of Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1274/2018
Record Dates: First submitted 2021-08-11; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Chronic Kidney Diseases; Malnutrition
Keywords: chronic kidney disease; Malnutrition
MeSH Terms: conditions — Renal Insufficiency, Chronic; Malnutrition

STUDY DESIGN:
Intervention Model Description: Participants were treated for six months with two different dietary prescriptions:
  1. LP group (n=17) was prescribed high calories/low proteins diet (30 Kcal/kg and 0.6-0.7gr/kg respectively). In order to assure prescribed calorie intake, this group was supplemented with commercial protein free products (protein content <2%).
  2. NP group (n=18) was prescribed high calories/normal proteins diet (30 kcal/kg and 0.8 gr/kg respectively).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LP group (Experimental): LP group (n=17) was prescribed high calories/low proteins diet (30 Kcal/kg and 0.6-0.7gr/kg respectively) supplemented with commercial protein free products (protein content <2%).
  Interventions: Dietary Supplement: LP group
- NP group (Active Comparator): NP group (n=18) was prescribed high calories/normal proteins diet (30 kcal/kg and 0.8 gr/kg respectively)
  Interventions: Other: NP group

INTERVENTIONS:
Dietary Supplement: LP group — LP group patients replaced pasta, bread, biscuits etc. with low protein substitutes. We allowed them to consume more animal products than NP, preferring white meat to red meat and trying to limit cold cuts as much as possible. Furthermore, they were advised to prefer fresh or frozen fish, instead of dried or smoked one as well as to prefer fresh cheeses to seasoned ones. As for legumes, we advised to combine them with bread or normal cereals, for protein complementarity.
  Arms: LP group
Other: NP group — NP group was given the indication to try to eat the second dish only once a day or to split the portion of the second plate between lunch and dinner, if they wanted to keep the habit of making the meal complete. It was also given the indication to prefer, among protein sources, those of plant origin. We also indicated to alternate or replace cow's milk with plant substitutes such as: rice, almonds' or oats' drinks. Furthermore, we suggested to prefer white meat and to avoid offal and processed meat. Moreover, we indicated to substitute dried or smoked fish with fresh or frozen one.
  Arms: NP group

SUMMARY:
It's a pilot study with an open label randomized-controlled design. Estimated number of patients should have been 38, taking in account of a maximal drop out up to 20% of the sample. We enrolled 35 patients, 27 of whom terminated the study as per protocol (14 in the Low protein (LP) group and 13 in the Normo Protein (NP) group).

Patients were treated for six months with two different dietary prescriptions:

1. LP group (n=17) was prescribed high calories/low proteins diet (30 Kcal/kg and 0.6-0.7gr/kg respectively). In order to assure prescribed calorie intake, this group was supplemented with commercial protein free products (protein content <2%).
2. NP group (n=18) was prescribed high calories/normal proteins diet (30 kcal/kg and 0.8 gr/kg respectively).

The primary hypothesis of the study was that in CKD patients at risk of malnutrition (4 ≤ MIS ≥7) with a persistent spontaneous low protein and calories intake, the prescription of a LP diet was not inferior to NP diet regarding the development of malnutrition (i.e.MIS ≥ 8).

We also wanted to test whether in these patients, the prescription of a LP diet was superior to the NP comparator regarding the control of the metabolic complication of chronic kidney diseases (i.e hyperphosphatemia, inflammation and metabolic acidosis), the progression on dyna/sarcopenia, inflammation and possibly on the progression of renal disease itself.

DETAILED DESCRIPTION:
Nutritional status will be evaluated through:

* Malnutrition Inflammation Score (MIS),
* Anthropometric measurements,
* albumin, prealbumin, transferrin,
* 24h urinary nitrogen,
* bioimpedance analysis (BIA),
* periodic 24h dietary diaries,
* International Society of Renal Nutrition and Metabolism (ISRNM),

Physical performance will be evaluated through:

* Short Physical Performance Battery (SPPB)
* Handgrip strength

Inflammation assessment:

* c-reactive protein (CRP)
* Interleukine-6 (IL6)
* whole blood Neutrophil/lymphocyte ratio

Renal function assessment:

* eGFR based on serum creatinine and cystatin C
* average creatinine and urea clearance

Uremic metabolic alteration:

* serum urea
* serum phosphate
* serum FGF23
* parathormone (PTH),
* plasma pH and bicarbonate

Time points of evaluation Dietary compliance has been assessed by a trained nutritionist at months 1, 2, 3 and 6. Dietary consumption was estimated by using dietary diaries and normalized catabolic protein rate (nPCR) measurement at baseline, 3 and at 6 months.

Nutritional status and physical performance have been evaluated monthly for the first three months and then at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* advanced CKD not yet on renal replacement therapy (10< - eGFRcreat <30 ml/min)
* age >65 years
* at risk of malnutrition at Malnutrition Inflammation Score (4≤MIS≤7)
* spontaneous low protein-energy intake (proteins < 0.8g/kg and energy < 25 kcal/kg).

Exclusion Criteria:

* Active chronic infectious diseases
* Heart failure of severity > NYHA2
* Active neoplastic diseases
* Inability to cooperate
* Presumed overall life expectancy < 6 month
* Decompensated liver diseases
* Malabsorption
* Decompensated thyroid o surrenal diseases
* Refusal to participate
* Immunosuppressive and/or steroid therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline MIS at 6th month | measured at baseline and 6 months.
  Malnutrition-inflammation score is a validated scoring system for the assessment of malnutrition and inflammation syndrome in patients with CKD. MIS involves the evaluation of ten different domains, each of which is categorized with 4 severity levels (score scale 0-3). A total score of 4-7 was considered indicative of mild malnutrition and a score ≥8 of severe malnourishment
Change from baseline serum albumin at 6th month | measured at baseline and at 6 months.
  in g/dL
intergroup MIS comparison at 6 months | 6th month
  Malnutrition-inflammation score is a validated scoring system for the assessment of malnutrition and inflammation syndrome in patients with CKD. MIS involves the evaluation of ten different domains, each of which is categorized with 4 severity levels (score scale 0-3). A total score of 4-7 was considered indicative of mild malnutrition and a score ≥8 of severe malnourishment
Intergroup comparison of the number of patients that reached a MIS ≥8 at 6 months | 6th month
  Malnutrition-inflammation score is a validated scoring system for the assessment of malnutrition and inflammation syndrome in patients with CKD. MIS involves the evaluation of ten different domains, each of which is categorized with 4 severity levels (score scale 0-3). A total score of 4-7 was considered indicative of mild malnutrition and a score ≥8 of severe malnourishment

SECONDARY OUTCOMES:
Differences of GFR estimated with creatinine | measured at baseline and at 6 months.
  In ml/min/1,73m^2
Differences of GFR estimated with cystatin C | measured at baseline and at 6 months.
  in ml/min/1,73m^2
Differences in serum urea | measured at baseline and at 6 months.
  in mg/dl
Differences in creatinine clarance | measured at baseline and at 6 months.
  in ml/min
Differences in phosphorous | measured at baseline and at 6 months.
  in mg/dl
Differences in FGF23 intact | measured at baseline and at 6 months.
  in pg/mL
Differences in FGF23 c-terminal | measured at baseline and at 6 months.
  in RU/mL
Differences in urinary phosphorous | measured at baseline and at 6 months.
  in mg/24h
Differences in PTH | measured at baseline and at 6 months.
  in ng/L
Differences in bicarbonate | measured at baseline and at 6 months.
  in mEq/L
Differences in pH | measured at baseline and at 6 months.
  pH
Differences in CRP | measured at baseline and at 6 months.
  in mg/dl
Differences in IL6 | measured at baseline and at 6 months.
  in pg/mL
Differences in the short physical performance battery scores | at months 1 and 6
  SPPB includes: test of standing balance, 4-meter walk and time to rise from a chair five times. Each SPPB component test is scored from 0 to 4. Higher scores indicate better physical performance
Differences of the handgrip strength | measured at baseline and at 6 months.
  in Kg. Handgrip strength was measured with Jamar dynamometer and was considered to be impaired for values <16kg in females and <27kg in males
Differences in the body composition (lean body mass, fat body mass, water) in the two study groups (bio impedance) | measured at baseline and at 6 months.
  water in L, Lean body mass in Kg/m2 and fat body mass in Kg/m2. Body composition was measured by using a multifrequency bioelectrical impedance analysis device (BCM- Body Composition Monitor, Fresenius Medical Care, Bad Homburg, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Simone Vettoretti, Dr, Principal Investigator — Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico di Milano, Milan, Italy
Locations (1):
- Unit of nephrology, dialysis and renal transplantation - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
since it is a collaborative study, the data may be made available to other researchers only following a specific and motivated request that must be approved by all members of the consortium

REFERENCES:
- [Background] Ikizler TA, Greene JH, Wingard RL, Parker RA, Hakim RM. Spontaneous dietary protein intake during progression of chronic renal failure. J Am Soc Nephrol. 1995 Nov;6(5):1386-91. doi: 10.1681/ASN.V651386. PMID 8589313
- [Background] Mitch WE. Malnutrition: a frequent misdiagnosis for hemodialysis patients. J Clin Invest. 2002 Aug;110(4):437-9. doi: 10.1172/JCI16494. No abstract available. PMID 12189236
- [Background] Mitch WE. Cachexia in chronic kidney disease: a link to defective central nervous system control of appetite. J Clin Invest. 2005 Jun;115(6):1476-8. doi: 10.1172/JCI25255. PMID 15931387
- [Background] Tom K, Young VR, Chapman T, Masud T, Akpele L, Maroni BJ. Long-term adaptive responses to dietary protein restriction in chronic renal failure. Am J Physiol. 1995 Apr;268(4 Pt 1):E668-77. doi: 10.1152/ajpendo.1995.268.4.E668. PMID 7733266
- [Background] Masud T, Young VR, Chapman T, Maroni BJ. Adaptive responses to very low protein diets: the first comparison of ketoacids to essential amino acids. Kidney Int. 1994 Apr;45(4):1182-92. doi: 10.1038/ki.1994.157. PMID 8007590
- [Background] Goodship TH, Mitch WE, Hoerr RA, Wagner DA, Steinman TI, Young VR. Adaptation to low-protein diets in renal failure: leucine turnover and nitrogen balance. J Am Soc Nephrol. 1990 Jul;1(1):66-75. doi: 10.1681/ASN.V1166. PMID 2104252
- [Background] Kopple JD, Monteon FJ, Shaib JK. Effect of energy intake on nitrogen metabolism in nondialyzed patients with chronic renal failure. Kidney Int. 1986 Mar;29(3):734-42. doi: 10.1038/ki.1986.59. PMID 3702224
- [Background] Garibotto G, Sofia A, Parodi EL, Ansaldo F, Bonanni A, Picciotto D, Signori A, Vettore M, Tessari P, Verzola D. Effects of Low-Protein, and Supplemented Very Low-Protein Diets, on Muscle Protein Turnover in Patients With CKD. Kidney Int Rep. 2018 Jan 11;3(3):701-710. doi: 10.1016/j.ekir.2018.01.003. eCollection 2018 May. PMID 29854979
- [Background] Ikizler TA, Burrowes JD, Byham-Gray LD, Campbell KL, Carrero JJ, Chan W, Fouque D, Friedman AN, Ghaddar S, Goldstein-Fuchs DJ, Kaysen GA, Kopple JD, Teta D, Yee-Moon Wang A, Cuppari L. KDOQI Clinical Practice Guideline for Nutrition in CKD: 2020 Update. Am J Kidney Dis. 2020 Sep;76(3 Suppl 1):S1-S107. doi: 10.1053/j.ajkd.2020.05.006. PMID 32829751
- [Background] Farrington K, Covic A, Aucella F, Clyne N, de Vos L, Findlay A, Fouque D, Grodzicki T, Iyasere O, Jager KJ, Joosten H, Macias JF, Mooney A, Nitsch D, Stryckers M, Taal M, Tattersall J, Van Asselt D, Van den Noortgate N, Nistor I, Van Biesen W; ERBP guideline development group. Clinical Practice Guideline on management of older patients with chronic kidney disease stage 3b or higher (eGFR <45 mL/min/1.73 m2). Nephrol Dial Transplant. 2016 Nov;31(suppl 2):ii1-ii66. doi: 10.1093/ndt/gfw356. No abstract available. PMID 27807144
- [Background] Rhee CM, Ahmadi SF, Kovesdy CP, Kalantar-Zadeh K. Low-protein diet for conservative management of chronic kidney disease: a systematic review and meta-analysis of controlled trials. J Cachexia Sarcopenia Muscle. 2018 Apr;9(2):235-245. doi: 10.1002/jcsm.12264. Epub 2017 Nov 2. PMID 29094800
- [Background] Fouque D, Kalantar-Zadeh K, Kopple J, Cano N, Chauveau P, Cuppari L, Franch H, Guarnieri G, Ikizler TA, Kaysen G, Lindholm B, Massy Z, Mitch W, Pineda E, Stenvinkel P, Trevino-Becerra A, Wanner C. A proposed nomenclature and diagnostic criteria for protein-energy wasting in acute and chronic kidney disease. Kidney Int. 2008 Feb;73(4):391-8. doi: 10.1038/sj.ki.5002585. Epub 2007 Dec 19. PMID 18094682
- [Result] Cupisti A, Brunori G, Di Iorio BR, D'Alessandro C, Pasticci F, Cosola C, Bellizzi V, Bolasco P, Capitanini A, Fantuzzi AL, Gennari A, Piccoli GB, Quintaliani G, Salomone M, Sandrini M, Santoro D, Babini P, Fiaccadori E, Gambaro G, Garibotto G, Gregorini M, Mandreoli M, Minutolo R, Cancarini G, Conte G, Locatelli F, Gesualdo L. Nutritional treatment of advanced CKD: twenty consensus statements. J Nephrol. 2018 Aug;31(4):457-473. doi: 10.1007/s40620-018-0497-z. Epub 2018 May 24. PMID 29797247
- [Result] Hanna RM, Ghobry L, Wassef O, Rhee CM, Kalantar-Zadeh K. A Practical Approach to Nutrition, Protein-Energy Wasting, Sarcopenia, and Cachexia in Patients with Chronic Kidney Disease. Blood Purif. 2020;49(1-2):202-211. doi: 10.1159/000504240. Epub 2019 Dec 18. PMID 31851983
- [Result] Deer RR, Volpi E. Protein Requirements in Critically Ill Older Adults. Nutrients. 2018 Mar 20;10(3):378. doi: 10.3390/nu10030378. PMID 29558388
- [Result] Cocks K, Torgerson DJ. Sample size calculations for pilot randomized trials: a confidence interval approach. J Clin Epidemiol. 2013 Feb;66(2):197-201. doi: 10.1016/j.jclinepi.2012.09.002. Epub 2012 Nov 27. PMID 23195919
- [Result] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Result] Vettoretti S, Caldiroli L, Armelloni S, Ferrari C, Cesari M, Messa P. Sarcopenia is Associated with Malnutrition but Not with Systemic Inflammation in Older Persons with Advanced CKD. Nutrients. 2019 Jun 19;11(6):1378. doi: 10.3390/nu11061378. PMID 31248132
- [Result] Afsar B, Sezer S, Ozdemir FN, Celik H, Elsurer R, Haberal M. Malnutrition-inflammation score is a useful tool in peritoneal dialysis patients. Perit Dial Int. 2006 Nov-Dec;26(6):705-11. PMID 17047239
- [Result] Maroni BJ, Steinman TI, Mitch WE. A method for estimating nitrogen intake of patients with chronic renal failure. Kidney Int. 1985 Jan;27(1):58-65. doi: 10.1038/ki.1985.10. PMID 3981873
- [Result] Legrand D, Vaes B, Mathei C, Adriaensen W, Van Pottelbergh G, Degryse JM. Muscle strength and physical performance as predictors of mortality, hospitalization, and disability in the oldest old. J Am Geriatr Soc. 2014 Jun;62(6):1030-8. doi: 10.1111/jgs.12840. Epub 2014 May 6. PMID 24802886
- [Result] Treacy D, Hassett L. The Short Physical Performance Battery. J Physiother. 2018 Jan;64(1):61. doi: 10.1016/j.jphys.2017.04.002. Epub 2017 Jun 20. No abstract available. PMID 28645532
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Result] Lau WL, Obi Y, Kalantar-Zadeh K. Parathyroidectomy in the Management of Secondary Hyperparathyroidism. Clin J Am Soc Nephrol. 2018 Jun 7;13(6):952-961. doi: 10.2215/CJN.10390917. Epub 2018 Mar 9. PMID 29523679
- [Result] Darmon P, Kaiser MJ, Bauer JM, Sieber CC, Pichard C. Restrictive diets in the elderly: never say never again? Clin Nutr. 2010 Apr;29(2):170-4. doi: 10.1016/j.clnu.2009.11.002. Epub 2009 Nov 22. PMID 19932533
- [Result] Wolfe RR, Miller SL, Miller KB. Optimal protein intake in the elderly. Clin Nutr. 2008 Oct;27(5):675-84. doi: 10.1016/j.clnu.2008.06.008. Epub 2008 Sep 25. PMID 18819733
- [Derived] Caldiroli L, Vettoretti S, Armelloni S, Mattinzoli D, Ikehata M, Molinari P, Alfieri C, Messa P, Castellano G. Possible Benefits of a Low Protein Diet in Older Patients With CKD at Risk of Malnutrition: A Pilot Randomized Controlled Trial. Front Nutr. 2022 Jan 26;8:782499. doi: 10.3389/fnut.2021.782499. eCollection 2021. PMID 35198584